CLINICAL TRIAL: NCT03160326
Title: The Quantitative Ultrasound Assessment of Lean and Intramuscular Adipose Tissue in Veterans With Chronic Kidney Disease
Brief Title: The QUALITY Vets Project: Muscle Quality and Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: AM-251-12-11-2015
Record Dates: First submitted 2016-10-05; First posted 2017-05-19 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Chronic Kidney Disease; Sarcopenia
Keywords: chronic kidney disease; ultrasound; muscle loss
MeSH Terms: conditions — Renal Insufficiency, Chronic; Sarcopenia; Muscular Atrophy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Currently there is no standard way to detect age-related skeletal muscle loss in patients with chronic kidney disease. Investigators are working on finding rapid and inexpensive ways to measure muscle size and fat within the muscle.

DETAILED DESCRIPTION:
The accelerated muscle wasting associated with chronic kidney disease (CKD) is a source of morbidity and an increased incidence of bone fracture secondary to falls. However, sarcopenia secondary to CKD is not routinely screened or assessed in this patient population. This protocol, "Quantitative Ultrasound Assessment of Lean and Intramuscular Adipose Tissue in Veterans Project" (i.e., QUALITY VETS) is a VA Center for Innovation (VACI) funded pilot study with the purpose of using a clinically viable sarcopenia screening approach for Veterans with CKD who are currently receiving care at the Renal Service.

The investigative team will screen and assess diminished muscle mass, quality, and performance in Veterans with CKD (Stage 3 and 4), and also examine the relationship between the muscle characteristics and estimated fall risk within the sample. Key outcome measures will be obtained within the domains of muscle performance (peak grip strength), functional status (Short Physical Performance Battery), estimates of tissue/body composition (diagnostic ultrasound and DXA), and fall risk (Timed Up-and-Go test). Secondary measures will include questionnaires regarding of fall avoidance, physical activity, depression, and quality of life (QoL).

The general analysis approach will be to characterize the proportion of participants with: sarcopenia based on the European Working Group on Sarcopenia in Older People (EWGSOP) algorithm, low muscle quality based on preliminary echogenicity cut off values and criterion strength values, and an elevated risk of falling based on the Timed Up-and-Go age-dependent cut off values. Investigators will determine the magnitude of association between the skeletal muscle outcomes and fall risk within the participant sample. Hazard ratios will be used to estimate the impact of the sarcopenia classification and echogenicity values on the positive classification of fall risk.

The optimal treatment of Veterans with CKD who have an elevated risk of falls may be enhanced by the timely identification of accelerated muscle changes. The QUALITY-VETS Project will help to determine appropriate screening and assessment strategies that could be implemented in subsequent longitudinal studies involving exercise interventions and fall prevention training.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients (with or without a gait aid)
* 18-84.9 years of age with CKD stage 3 or 4
* Receiving care at the DC or SF VA Medical Center Renal Service
* Able to speak and read English
* Orientation to person, place, and time

Exclusion Criteria:

* Acute renal failure
* Pregnancy
* Any uncontrolled cardiovascular or musculoskeletal disease that, in the opinion of the principal investigator, could make participation unsafe
* Body size exceeds the dimensional limits of the DXA scanner

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participating Veterans in this study will undergo their standard examination by the DC or SF VA Medical Center Renal Service staff physicians and will be formally staged for CKD. Fifty adult patients with Stage 3 or 4 CKD (i.e., a definitive CKD diagnosis, but prior to the need for dialysis) will be enrolled following consent and then scheduled for the study assessments at their local study center.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-10 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Muscle Quality | day 1
  Muscle measurements at 6 sites using diagnostic ultrasound (grayscale levels, 0-255)
Lean Body Mass | day 1
  Dual Energy X-ray Absorptiometry (DXA) scan (kg/m2)
Grip Strength | day 1
  Measured using a dynamometer (kg)
Short Physical Performance Battery | day 1
  Performance-based functional assessment battery; scores range from 0 (worst performance) to 12 (best performance)
Timed Up-and-Go | day 1
  Performance-based fall risk assessment

SECONDARY OUTCOMES:
Height | day 1
  Participant height in meters
Weight | day 1
  Participant weight in kilograms
Hip/waist circumference | day 1
  Participant hip and waist circumference in centimeters
Body composition | day 1
  Body composition data in presented in percentages of the body composed of water, bone, muscle, and fat using a bioelectric scale
Isometric peak knee extension force | day 1
  Measured using a load cell
Activities-Specific Balance Confidence Scale | day 1
  Mobility questionnaire
SF-36 - Physical Function Scale | day 1
  General physical functioning questionnaire
Falls Efficacy Scale | day 1
  Fall avoidance behavior questionnaire
Physical Activity Scale for the Elderly | day 1
  Self-reported estimate physical activity
Sarcopenia-specific QoL scale (SarQoL) | day 1
  Self-reported health-related quality of life
CES-D | day 1
  Depression Scale

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Delgado, MD, Principal Investigator — San Francisco VA Medical Center
Locations (2):
- United States (2):
  - San Francisco VA Medical Center, San Francisco, California
  - Washington DC VA Medical Center, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared between the two study sites: the Washington DC and San Francisco VA Medical Centers

REFERENCES:
- [Derived] Gollie JM, Harris-Love MO, Patel SS, Shara NM, Blackman MR. Rate of Force Development Is Related to Maximal Force and Sit-to-Stand Performance in Men With Stages 3b and 4 Chronic Kidney Disease. Front Rehabil Sci. 2021 Sep 28;2:734705. doi: 10.3389/fresc.2021.734705. PMID 34708217